CLINICAL TRIAL: NCT06095050
Title: Efficacy of Lipiodol Embolization for Chronic Tendinopathy of the Rotator Cuff
Brief Title: Embolization Treatment of Chronic Refractory Shoulder Tendinopathy
Acronym: ELECTRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Yan Epelboym, M.D.,M.P.H., Interventional Radiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P002574
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Shoulder Pain; Tendinopathy; Rotator Cuff Tendinitis; Rotator Cuff Tendinosis; Embolization; Arterial Occlusion
Keywords: pain; shoulder pain; tendinopathy
MeSH Terms: conditions — Shoulder Pain; Tendinopathy; Rotator Cuff Injuries; Arterial Occlusive Diseases; Pain | interventions — Embolization, Therapeutic; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Single center prospective randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Embolization (Experimental): Angiography will be performed to identify hyperemic neovasculature arising from one or more of branch shoulder arteries. After localizing the abnormal neovessels a microcatheter will be inserted coaxially and selectively placed in the targeted artery(ies). The abnormal vessels will be embolized with Lipiodol emulsion (Guerbet, Villepinte, France) The embolic agent will be used under an investigational device exemption from the FDA. The embolic will be injected in small volume increments until blood flow stagnates in the target artery(ies).
  Angiography and embolization will be repeated until the hyperemia is markedly reduced as demonstrated on digital subtraction angiography.
  Subjects will participate in structured physical therapy consisting of 3 months of eccentric strength training. This twelve-week program will consist of 4 PT sessions at week 0, week 4, week 8, and week 12.
  Interventions: Device: Embolization; Other: Physical Therapy
- Physical Therapy (Active Comparator): Subjects will participate in structured physical therapy consisting of 3 months of eccentric strength training. This twelve-week program will consist of 4 PT sessions at week 0, week 4, week 8, and week 12.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Device: Embolization — Superselective arterial embolization of hyperemic vasculature in the symptomatic shoulder (utilizing the IDE approved device: Lipiodol) followed by structured physical therapy sessions.
  Arms: Embolization
Other: Physical Therapy — Subjects will participate in structured physical therapy consisting of 3 months of eccentric strength training. This twelve-week program will consist of 4 PT sessions at week 0, week 4, week 8, and week 12.

SUMMARY:
This is a randomized controlled trial in which patients with moderate to severe shoulder pain (Visual Analog Scale (VAS) > 40), in the setting of rotator cuff tendinopathy refractory to conservative treatment, will be enrolled.

The primary aim of the study is to estimate the effect of transcatheter arterial embolization (TAE) with physical therapy (PT) vs PT alone on the change in shoulder pain at 12-month follow up. Scientific objectives also include an assessment of safety of the intervention, assessment of changes in Patient-Reported Outcomes Measurement Information System (PROMIS) Upper Extremity score, Shoulder Pain and Disability Index (SPADI) scores, MRI Tendinopathy Score between the TAE + PT and PT groups.

DETAILED DESCRIPTION:
This is a single center prospective randomized controlled study at Brigham & Women's Hospital (BWH), a teaching hospital of Harvard Medical School. Patients with clinical and MRI findings of shoulder tendinopathy, moderate to severe shoulder pain (VAS > 40), and pain refractory to at least 6 months of physician directed conservative therapy will be eligible for enrollment.At screening patient will undergo a shoulder MRI to evaluate for tendinopathy, and patients with complete full thickness tendon tears will be excluded.

Patients will be randomized to either the TAE +PT or PT group. Patients in the TAE + PT group will undergo angiography to evaluate branch shoulder arteries for hyperemia. If hyperemia is present, then embolization will be performed. This treatment will be followed by 3 months of structured PT. Patients in the PT group will undergo 3-months of structured physical therapy with isolated eccentric exercises.

ELIGIBILITY:
Inclusion Criteria:

1. Male, female, transgender female, transgender male, non-binary
2. Moderate to severe shoulder pain (VAS > 40)
3. Pain refractory to at least 6 months of physician-directed conservative therapy (analgesics or injections or PT), including a minimum of 6 weeks of PT
4. Willing, able, and mentally competent to provide informed consent and to tolerate angiography and physical therapy

Exclusion Criteria:

1. History of peripheral arterial disease or peripheral artery disease symptoms including claudication, diminished or absent upper/lower extremity pulses, or known upper extremity arterial atherosclerosis or occlusion that would limit selective angiography
2. Known history of anaphylaxis to iodinated contrast agents or gadolinium based contrast
3. Acute kidney injury
4. Allergy to poppy seeds or lipiodol
5. Renal dysfunction as defined by serum creatinine >1.6 dl/mg or eGFR <60 obtained within 30 days of procedure.
6. Uncorrectable coagulopathy (platelet count < 50,000, international normalized ratio >1.8 within 30 days of procedure
7. Active systemic or local upper extremity infection
8. Patient pregnant, intending to become pregnant during the study.
9. Prior shoulder replacement surgery
10. Prior rotator cuff repair surgery
11. Previous history of complete full-thickness tear of the rotator cuff
12. Presence of non-MRI compatible devices (e.g., non-compatible cardiac pacemaker).

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-01-16 (Estimated); Study Completion 2028-04-21 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale Pain (VAS) Score | 12 months
  The difference in shoulder visual analog pain scale scores between TAE +PT and PT groups obtained 12 months following intervention vs. pre-intervention. The visual analog scale is ratio scale from 0 to 100 which measures pain symptoms. On this scale higher numbers indicated more severe pain symptoms.

SECONDARY OUTCOMES:
Adverse Events | 12 months
  Compare the safety of TAE + PT relative to PT by recording adverse events at 1 month, 3 months, 6 months, and 12 months post intervention
Patient-Reported Outcomes Measurement Information System Upper Extremity | 12 months
  Estimate the effect of TAE + PT vs PT on the change in Patient-Reported Outcomes Measurement Information System Upper Extremity scores at 1, 3, 6 and 12-months. A higher score indicates a better outcome. The scores can range from 15 to 61and are scored on what is called a T-score, a metric which reflects one standard deviation for each 10 points.
Shoulder Pain and Disability Index | 12 months
  estimate the effect of TAE + PT vs PT on the change in Shoulder Pain and Disability Index scores at 1, 3, 6 and 12-months. The scale is a ratio scale of 0 to 130 with higher scores indicating greater degree of pain and disability.
MRI Tendinopathy scores | 12 months
  Estimate the effect of TAE + PT vs PT on the change in MRI Tendinopathy scores at baseline and 12-months. The scale is ordinal and ranges from 0 to 3 with higher scores indicating a greater degree of tendinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Epelboym, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States